Informed consent for participation in the clinial trial

## Peripheral nerveblocks for reduction of distal forearm fractures

Declaration from trial participant

I have received both oral and written information and I know enough about aims, methods, gains and benefits of the trial to accept participation.

I know that participation is **voluntary** and that I may retract my consent at any given time without losing any current or future rights to treatment.

I give my consent to trial participation and have been given a copy of this informed consent form as well as a copy of the written trial information for my own use.

| Participant nar | e: |
|---|---|
| Date: | Signature: |
| Do you wish t<br>treatment? | receive information on the results of the trial and any impact it may have had on you |
| Yes | ick X) No(tick X) |
| Declaration fro | n physician delivering information |
| declare that t | e trial participant has received both oral and written trial information. |
| n my conviction | sufficient information has been given to obtain an informed consent for trial participation. |
| Name of physi | an delivering information: |
| Date: | Signature: |
| Project identif | ation numbers: |
| | anish Data Protection Agency: 1-16-02-875-17 |
| | he Central Denmark Region Committees on Health Research Ethics: 1-10-72-210-17 |